CLINICAL TRIAL: NCT03009422
Title: Fractional CO2 Laser With Topical Pentostam Treatment for Cutaneous Leishmaniasis.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TASMC-14-OA-371-CTIL
Record Dates: First submitted 2016-12-14; First posted 2017-01-04 (Estimated); Last update posted 2017-01-04 (Estimated); Status verified 2016-12

CONDITIONS: Leishmaniasis
MeSH Terms: conditions — Leishmaniasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment (Experimental): CO2 fractional laser with local application of Pentostam
  Interventions: Drug: Local application pentostam; Device: fractional CO2 laser
- control (Active Comparator): Intra-lesinal Pentostam injedction
  Interventions: Drug: intra-lisional pentostam

INTERVENTIONS:
Drug: Local application pentostam
  Arms: Treatment
Drug: intra-lisional pentostam
  Arms: control
Device: fractional CO2 laser
  Arms: Treatment

SUMMARY:
The investigators will compare the common treatment for cutaneous leishmaniasis with intra-lesional Pentostam to fractional CO2 laser with topical application of Pentostam.

Outcome will be final scar appearance assesd by two dermatologist and pain measurement by VAS.

DETAILED DESCRIPTION:
20 healthy patients diagnosed will cutaneous leishmaniasis with more than one lesion will be recruited.

Half of the lesions will be treated with intra-lesional injections of Pentostam, and the other half by CO2 laser with topical application of Pentostam.

Each lesion will recieve 3 treatments, one month apart between treatments. The patients will scale pain level of each treatment. Final scar appearance will be assessed by two dermatologists, without knowing what treatment was applied to each lesion.

ELIGIBILITY:
Inclusion Criteria:

* Objective cutaneous leishmaniasis diagnosis.
* More than one Lesion

Exclusion Criteria:

* Previous treatment
* Abnormal scarring

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2014-11; Primary Completion 2017-02 (Estimated); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
scar appearance | At sixth month
  Each lesion will be photographed prior to treatment and at 6th month (Three months after last (3rd) treatment).Two dermatologist will asses each lesion outcome

SECONDARY OUTCOMES:
Pain assessed by VAS | at one month, two months, and three months

REFERENCES:
- [Background] Monge-Maillo B, Lopez-Velez R. Therapeutic options for old world cutaneous leishmaniasis and new world cutaneous and mucocutaneous leishmaniasis. Drugs. 2013 Nov;73(17):1889-920. doi: 10.1007/s40265-013-0132-1. PMID 24170665
- [Background] Al-Natour SH. Update in the treatment of cutaneous leishmaniasis. J Family Community Med. 2009 May;16(2):41-7. PMID 23012189
- [Background] Arfan-ul-Bari, Simeen-ber-Rahman. Scar leishmaniasis. J Coll Physicians Surg Pak. 2006 Apr;16(4):294-5. PMID 16624197
- [Background] Kim DW, Hwang NH, Yoon ES, Dhong ES, Park SH. Outcomes of ablative fractional laser scar treatment. J Plast Surg Hand Surg. 2015 Apr;49(2):88-94. doi: 10.3109/2000656X.2014.919927. Epub 2014 May 21. PMID 24845386
- [Background] AlGhamdi K, Khurrum H. Successful treatment of atrophic facial leishmaniasis scars by co2 fractional laser. J Cutan Med Surg. 2014 Nov;18(6):379-84. doi: 10.2310/7750.2014.13175. PMID 25348758
- [Background] Sklar LR, Burnett CT, Waibel JS, Moy RL, Ozog DM. Laser assisted drug delivery: a review of an evolving technology. Lasers Surg Med. 2014 Apr;46(4):249-62. doi: 10.1002/lsm.22227. Epub 2014 Mar 24. PMID 24664987
- [Background] Bloom BS, Brauer JA, Geronemus RG. Ablative fractional resurfacing in topical drug delivery: an update and outlook. Dermatol Surg. 2013 Jun;39(6):839-48. doi: 10.1111/dsu.12111. Epub 2013 Jan 7. PMID 23294061